CLINICAL TRIAL: NCT02070003
Title: Perioperative Recovery of Moods, Opioids, and Pain Trial (PROMPT)
Acronym: PROMPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer Hah, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26234
Record Dates: First submitted 2014-02-10; First posted 2014-02-24 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Opioid Cessation
MeSH Terms: interventions — Motivational Interviewing

ARMS (2):
- Motivational Interviewing and Physician Guided Opioid Weaning (Experimental): Patients will go through motivational interviewing with the study physician via phone once a week for 7 weeks, and once a month up to a year as applicable, until patient completes the protocol.
  Interventions: Behavioral: Motivational Interviewing and Physician Guided Opioid Weaning
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Motivational Interviewing and Physician Guided Opioid Weaning
  Arms: Motivational Interviewing and Physician Guided Opioid Weaning

SUMMARY:
The investigators aim to characterize the relationship between changes in emotional distress, opioid use, and pain throughout surgery and recovery. Additionally, the investigators aim to compare the effectiveness of post-surgical motivational interviewing and physician-guided opioid weaning vs. usual care on reducing persistent opioid use. Overall, the proposed research will advance knowledge regarding the role of psychological factors contributing to persistent opioid use after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Undergoing a scheduled surgery
* English speaking
* Ability and willingness to complete questionnaires and assessments.

Exclusion Criteria:

* Any conditions causing inability to complete baseline, telephone and internet assessments (e.g. education, cognitive ability, mental status, medical status)at the discretion of the investigator.
* Known Pregnancy
* Elevated Suicidality as assessed by an answer of 2 or greater on question 9 of the Beck Depression Inventory assessing suicidal thoughts.
* Coexisting Chronic Pain Disorder of moderate severity in area other than surgical target

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-11-26 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Trial Feasibility - The proportion of people consented who complete the study in the group to which they were randomized | Duration of the study - up to 2 years per participant
  Factors that contribute to non-completion of the study, measured at baseline for each patient, will be analyzed.

SECONDARY OUTCOMES:
Efficacy - time to opioid cessation | Duration of the trial - Up to 2 years per participant
  Time to opioid cessation between the two groups will be analyzed using survival analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Hah, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

REFERENCES:
- [Derived] Hah JM, Trafton JA, Narasimhan B, Krishnamurthy P, Hilmoe H, Sharifzadeh Y, Huddleston JI, Amanatullah D, Maloney WJ, Goodman S, Carroll I, Mackey SC. Efficacy of motivational-interviewing and guided opioid tapering support for patients undergoing orthopedic surgery (MI-Opioid Taper): A prospective, assessor-blind, randomized controlled pilot trial. EClinicalMedicine. 2020 Oct 16;28:100596. doi: 10.1016/j.eclinm.2020.100596. eCollection 2020 Nov. PMID 33294812